CLINICAL TRIAL: NCT04289532
Title: First-in-human Pilot Study of an Integrin α6-targeted Radiotracer for SPECT Imaging of Breast Cancer
Brief Title: Integrin α6-targeted SPECT Imaging of Breast Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: China-Japan Union Hospital, Jilin University (Other); Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Fan Wang, Professor, Beijing University Health Science Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 010006
Record Dates: First submitted 2020-02-25; First posted 2020-02-28 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
Keywords: Breast cancer; integrin α6; SPECT
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 99mTc-RWY SPECT/CT (Experimental): Volunteers and patients were injected intravenously with 11.1 MBq/kg of 99mTc-RWY in one dose and underwent SPECT/CT scan 30-60 min later.
  Interventions: Drug: 99mTc-RWY

INTERVENTIONS:
Drug: 99mTc-RWY — 99mTc-RWY were injected into volunteers and patients before the SPECT/CT scans .
  Other Names: 99mTc-labeled peptide targeting integrin α6

SUMMARY:
A novel radiotracer 99mTc-RWY targeting Integrin α6 was developed, and the pilot first-in-human study for SPECT imaging of breast cancer was performed in seven healthy volunteers and two breast cancer patients to assess the safety and potential clinical applications of 99mTc-RWY.

DETAILED DESCRIPTION:
Integrin α6 associates with the survival and migration of breast cancer cells, which emerges as a predictor of reduced overall survival and worse prognosis. In this study, we developed an integrin α6-targeted radiotracer 99mTc-RWY for SPECT imaging of breast cancer. The safety, biodistribution and radiation dosimetry were studied in seven healthy volunteers, and the clinical potential of 99mTc-RWY was examined in two breast cancer patients. A single dose of 11.1 MBq/kg 99mTc-RWY was injected intravenously. Visual and semiquantitative methods were used to assess the SPECT/CT images. The routine Hematoxylin-Eosin (HE) staining and immunohistochemistry (IHC) staining were subsequently carried out to confirm the Integrin α6 expression of tumors.

ELIGIBILITY:
Inclusion criteria:

* Healthy volunteers.
* Body mass index (BMI) at 19 to 25 [Body mass index = body weight (kg)/ height squared (m2)];
* Clinical laboratory tests (heart, liver, kidney, blood) indicators are in the normal range or abnormalities without clinical significance;
* Informed written consents were obtained from all 9 subjects before the procedure.
* Patients in suspicion of breast cancer by mammography or ultrasonography, and being able to provide basic information.

Exclution Criteria:

• The investigator judged that it is not suitable for clinical trials based on the overall situation of the volunteers and patients.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Blood Clearance | 1,3,5,10,15,30,60,120 minutes post-injection
  The %ID (the radioactivity of the blood at each time period/the total injection activity) is calculated.
Excretion | 0-24 hours post-injection
  The %ID (the radioactivity of the urine at each time period/the total injection activity) is calculated.
Biodistribution | 0.5,1,2,4,24 hours post-injection
  Area under the activity-time curve from hour 0 to last measurable activity.
SPECT/CT imaging | post-injection
  Image brightness is observed。
Distributed in organs | 0.5,1,2,4,24 hours post-injection
  The %ID (the radioactivity of the main organs at each time period/the total injection activity) is calculated.

SECONDARY OUTCOMES:
Incidence of adverse events | 1 week post-injection
  Adverse events within 1 week after the injection and scanning were followed and assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Health Science Center, Beijing, Beijing Municipality, China